CLINICAL TRIAL: NCT06705192
Title: Open-label Multiple Dosing Study in Asymptomatic GRN-frontotemporal Dementia Patients to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VES001.
Brief Title: Study in Asymptomatic GRN-FTD Patients to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VES001
Acronym: SORT-IN-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mads Kjolby (Industry)
Responsible Party: Sponsor-Investigator, Mads Kjolby, Chief Medical Officer, Vesper Biotechnologies ApS
Organization: Vesper Biotechnologies ApS (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ph1b/FTD002; 2024-513258-31-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-22; First posted 2024-11-26 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Frontotemporal Dementia; Asymptomatic Condition
MeSH Terms: conditions — Dementia; Frontotemporal Dementia; Asymptomatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a single cohort, investigating 2 distinct dose levels (Dose 1: 360 mg and Dose 2: 900 mg) (Other): The study follows a MAD design within a single cohort, investigating 2 distinct dose levels (Dose 1: 360 mg and Dose 2: 900 mg), consecutively over a 3-month period.
  Dose 1 at 360 mg (2 capsules of 180 mg in the morning) Dose 2 at 900 mg (2 capsules of 180 mg in the morning [360 mg], 3 capsules of 180 mg in the evening [540 mg])
  Interventions: Drug: VES001

INTERVENTIONS:
Drug: VES001 — VES001 is an oral, blood brain barrier ligand of sortilin.
  VES001 will be administered orally as a solid within a gelatine capsule without excipients; the capsule strength will be 180 mg.

SUMMARY:
This is an open-label, multiple dosing study in asymptomatic GRN-FTD carriers to investigate the safety, tolerability, PK, and PD of VES001. The study follows a MAD design within a single cohort, investigating 2 distinct dose levels (Dose 1: 360 mg and Dose 2: 900 mg), consecutively over a 3-month period. A total of 6 participants will be recruited over a fixed enrolment period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Has provided signed informed consent, prior to any study-mandated procedure.
* Has a BMI of ≥ 18 to ≤ 32 kg/m2, and with a minimum weight of 50 kg
* Is an asymptomatic carrier of the GRN mutation, previously confirmed via genetic testing AND historical records (as documented by FRS and FTLD-CDR-NACC-SB) available for review by the investigator

Note: Genetic testing for GRN mutation status will not be conducted as part of methodology or procedures in this study. The study relies on the previously confirmed GRN mutation data in medical history of the potentially eligible participants.

* In good physical health assessed by the investigator and medical history of the participant, physical examinations (PEs), laboratory tests, ECGs, and vital signs
* Is a FOCBP; as defined in CTFG 2020, must have a negative urine pregnancy test at screening and agree to heterosexual abstinence or the use at least 1 highly effective form of contraception (with a failure rate of <1% per year when used consistently and correctly), from the start of the screening period through 90 days after the last dose of the study drug (Appendix 3). All females are considered of childbearing potential unless they are postmenopausal (at least 12 consecutive months of amenorrhea in the appropriate age group without other known or suspected cause) or have been sterilised surgically (e.g., hysterectomy, bilateral oophorectomy, bilateral salpingectomy).
* Is a male participant who has not had a vasectomy and is sexually active with FOCBP must agree to use a barrier method of birth control from the start of the screening period through 90 days after the last dose of the study drug
* Is a male participant who must agree not to donate sperm from the start of the screening period, through the study, and for at least 90 days after the last dose of the study drug
* Is a female participant who must agree not to donate ova from the start of the screening period, through the study, and for at least 90 days after the last dose of the study drug
* Has the ability to communicate well with the investigator in the Dutch language (at the Erasmus Medical Centre) or English language (at the UCL) and willing to comply with the study restrictions.

Exclusion Criteria:

* Has evidence of any active or chronic disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would pose an unacceptable risk to the participant in the opinion of the investigator (following a detailed medical history, physical examination, vital signs [SBP, DBP, HR, respiratory rate, body temperature], and 12-lead ECG). Minor deviations from the normal range may be accepted, if judged by the investigator to have no clinical relevance.
* Has a history of any known neurologic disease, cognitive impairment, diagnosed abnormal cognitive decline related to the participant's age, a history of seizure, or (significant) head trauma.
* Has a history of active malignancy within the last 5 years, with the exception of fully resected cell carcinoma of the skin.
* Has clinically significant abnormalities, as judged by the investigator, in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel, and urinalysis). In the case of uncertain or questionable results, tests performed during screening may be repeated before dosing to confirm eligibility or judged to be clinically irrelevant for healthy participants
* Tests positive for HBsAg, HCV Ab, HIV1 Ab, or HIV2 Ab at screening.
* Has SBP greater than 140 (untreated hypertension) or less than 90 mm Hg, and DBP greater than 90 or less than 50 mm Hg at screening.
* Has abnormal findings in the resting ECG at screening defined as:

  1. QTcF > 450 or < 300 msec for males and QTcF > 470 or < 300 msec for females
  2. Notable resting bradycardia (HR < 45 bpm) or tachycardia (HR > 100 bpm)
  3. Personal or family history of congenital long QT syndrome or sudden death attributed to underlying heart disease
  4. ECG with QRS and/or T-wave judged to be unfavorable for a consistently accurate QT measurement (e.g., neuromuscular artefact that cannot be readily eliminated, arrhythmias, indistinct QRS onset, low amplitude T-wave, merged T- and U-waves, prominent U-waves)
* Has evidence of atrial fibrillation, atrial flutter, complete branch block, Wolf-Parkinson-White Syndrome, or cardiac pacemaker
* Meets criteria that would preclude a LP, such as:

  1. a local infection at the site of the LP
  2. < 50 × 10E3/μL platelet count at screening
  3. clinically significant coagulation abnormality
  4. significant active bleeding, treatment with an anticoagulant, or treatment with 2 or more antiplatelet agents
  5. history of clinically significant back pathology and/or back injury (e.g., degenerative disease, spinal deformity, or spinal surgery) that may predispose to complications or technical difficulty with LP
* Has any confirmed significant allergic reactions (urticaria or anaphylaxis) against any drug, or multiple drug allergies (non-active hay fever is acceptable).
* Uses any medications (prescription or OTC), within 14 days of study drug administration, or less than 5 half-lives (whichever is longer). Exceptions are paracetamol (up to 4 g/day) and ibuprofen (up to 1.2 g/day).
* Uses any vitamin, mineral, herbal, and dietary supplements within 7 days of study drug administration, or less than 5 half-lives (whichever is longer).
* Participated in an investigational drug or device study (last dosing of previous study was within 90 days or less than 5 elimination half-lives of the investigational treatment, whichever is longer, before first dosing of this study).
* Has any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence, psychiatric disease, or usage of anti-psychotic medications.
* Has a history of abuse of addictive substances (alcohol, illegal substances, drug abuse, or regular user of sedatives, hypnotics, tranquillisers, or any other addictive agent) in the past 2 years.
* Tests positive for drugs of abuse at screening or Day 1.
* Is a smoker of more than 10 cigarettes per day prior to screening or who use tobacco products equivalent to more than 10 cigarettes per day and unable to abstain from smoking while in the unit.
* Is demonstrating excess in caffeine consumption (more than 8 cups of coffee or equivalent per day)
* Has had a loss or donation of blood over 500 mL within 3 months (males) or 4 months (females) prior to screening or intention to donate blood or blood products during the study.
* Is a female, who is pregnant, breast-feeding, or planning to become pregnant during the study.
* Has any surgical or medical condition possibly affecting drug absorption (e.g., gastrectomy).
* Is, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide.
* Has answered "yes" to either Question 4 or Question 5 on the "Suicidal Ideation" portion of the C-SSRS and the ideation occurred within the past 6 months OR has answered "yes" to any of the suicide-related behaviours on the "Suicidal Behaviour" portion of the C-SSRS and the behaviour occurred within the past 1 year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-05 (Actual)

PRIMARY OUTCOMES:
Change in PGRN levels in CSF at Day 28 and Day 84 compared to baseline | 16 weeks
  Three (3) CSF samples will be obtained The total amount of CSF collected from each participant over the duration of the study, will not exceed 55 mL.
Change in PGRN levels in plasma at Day 28 and Day 84 compared to baseline | 16 weeks
  PD samples will be obtained 32 times

SECONDARY OUTCOMES:
To evaluate the CSF PK profile of VES001 following multiple oral doses in asymptomatic GRN-FTD carriers | 16 weeks
  Two (2) CSF PK parameters: Cmax will be obtained
To evaluate the CSF PK profile of VES001 following multiple oral doses in asymptomatic GRN-FTD carriers | 16 weeks
  Two (2) CSF PK parameters: tmax will be obtained
To evaluate the CSF PK profile of VES001 following multiple oral doses in asymptomatic GRN-FTD carriers | 16 weeks
  Two (2) CSF PK parameters: t1/2, will be obtained
To evaluate the CSF PK profile of VES001 following multiple oral doses in asymptomatic GRN-FTD carriers | 16 weeks
  Two (2) CSF PK parameters: Vz/F will be obtained
To evaluate the CSF PK profile of VES001 following multiple oral doses in asymptomatic GRN-FTD carriers | 16 weeks
  Two (2) CSF PK parameters: CL/F will be obtained
To evaluate the concentration of VES001 in CSF in all participants compared to baseline | 16 weeks
  Three (3) CSF samples will be obtained and analysis will be performed at D28 and Day 84 compared to baseline
To evaluate the concentration of VES001 in plasma/CSF ratio in all participants compared to baseline | 16 weeks
  Three (3) CSF samples will be obtained and analysis will be performed at D28 and Day 84 compared to baseline
All participants with treatment-related adverse events as assesed by CTCAE v 4.0 will be evaluated | 16 weeks
  Safety and tolerability including the severity and incidence of TEAEs, SAEs, and SUSARs of all participants will be assessed by the following endpoints: Monitoring and recording of AEs, SAEs, and SUSARs.
  For all safety assessments, the investigator will determine whether the results are clinically significant, which is defined as any variation in a result that has medical relevance and may result in an alteration in medical care (e.g., active observation, diagnostic measures, or therapeutic measures). If clinical significance is noted, the result and reason for significance will be documented and an AE reported on the AE page of the participant's eCRF. The investigator will monitor the participant until the result has reached the reference range or the result at Screening, or until the investigator determines that FU is no longer medically necessary.
To evaluate the safety and tolerability of clinical laboratory test results following multiple oral doses of VES001 in asymptomatic GRN-FTD carriers | 16 weeks
  All participants will be assessed by following endpoint; Severity and incidence of clinical laboratory test results. Clinical laboratory tests will be performed by the local site laboratories at UCL and Erasmus Medical Center. Blood and urine samples will be collected under fasting conditions (not eat or drink anything other than water for at least 4 hours before sample collections) and will be prepared using standard procedures. Measurements will be completed before VES001 dosing at all onsite visit with a total of eight (8) examinations.
  Repeat clinical laboratory tests may be performed at the discretion of the investigator, if necessary, to evaluate inclusion and exclusion criteria or clinical laboratory abnormalities. The clinical laboratory that will perform the tests will provide the reference ranges for all clinical laboratory parameters.
Evaluation of safety and tolerability of 12-lead ECG results & vital signs measurements following multiple oral doses of VES001 in asymptomatic GRN-FTD carriers | 16 weeks
  All participants will be assesed by following endpoints; changes in vital sign measurements and 12-lead ECG results; Vital signs will be measured within 15 minutes before and after VES001 dosing and will include SBP and DBP, heart rate, respiratory rate, and body temperature.
  Single 12-lead ECG will be performed within 15 minutes before and after VES001 dosing (assessments will include comments on whether the tracings are normal or abnormal, rhythm, presence of arrhythmia or conduction defects, morphology, any evidence of myocardial infarction, or ST-segment, T-wave, and U-wave abnormalities. In addition, measurements of the following intervals will be measured and reported: RR interval, PR interval, QRS width, QT interval, and QTcB and QTcF intervals).
Evaluation of safety and tolerability of physical/neurological examination findings and C-SSRS questionnaire findings following multiple oral doses of VES001 in asymptomatic GRN-FTD carriers | 16 weeks
  All participants will be assessed by following endpoints:
  A full physical and neurological examination will be performed at Screening (at minimum, assessment of the skin, head, ears, eyes, nose, throat, neck, thyroid, lungs, heart, abdomen, lymph nodes, cardiovascular and musculoskeletal system/extremities). Only targeted physical and neurological examination will be performed after Screening visit. Height and weight will be measured, and BMI calculated at Screening only. Only weight will be measured, and BMI calculated at the FU/EOS visit.
  The C-SSRS is a series of questions to assess suicidal ideation and behavior. Because the effect of VES001 occurs within the CNS, participants will be needed to complete a paper-based C-SSRS to collect data and monitor suicidal ideation and intent at the specified twelve (12) time points.
  Unscheduled assessments may be performed if any relevant AE is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mads Kjoelby, MD, PhD, Principal Investigator — Vesper Bio
Locations (2):
- Erasmus University Medical Center, Rotterdam, Netherlands
- Leonard Wolfson Experimental Neurology Centre CRF National Hospital for Neurology and Neurosurgery, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No